CLINICAL TRIAL: NCT06062342
Title: Five Point Initiative: A Cluster Randomized Trial of a Bundled Implementation Strategy to Address the HIV Epidemic in Black Communities
Brief Title: Five Point Initiative: A Bundled Implementation Strategy to Address the HIV Epidemic in Black Communities
Acronym: FPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sannisha K Dale, Associate Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20230484; 1R01MH134269-01 (NIH)
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hiv
Keywords: HIV prevention; HIV testing; PrEP; Implementation Science
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge trial and all zip codes cross over from pre-assessment period (control) to active intervention. The time/order in which zip codes enter the stepped wedge is the unity of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FPI Group (Experimental): Participants in this group will receive the FPI intervention at any FPI coordinated outreach event (4-5 hours) during a 21 month period
  Interventions: Behavioral: FPI
- Pre-intervention Assessment Group (No Intervention): We will conduct pre-assessment events (4-5 hours) during 1.5 months in each zip code (prior to the introduction of the FPI intervention) to capture information from residents /participants via survey.

INTERVENTIONS:
Behavioral: FPI — The FPI intervention will be conducted twice per month (across 21 months) in a zip code, and each event will last approximately 4-5 hours. At the event, participants will receive HIV testing, PrEP linkage (e.g., prescription) and knowledge, and condom and use/access.
  Arms: FPI Group

SUMMARY:
The purpose of this study is to assess the effectiveness of the FPI bundled implementation strategy in increasing HIV testing, Pre-exposure prophylaxis (PrEP) linkage (e.g., prescription) and knowledge, and condom use/access.

ELIGIBILITY:
Inclusion Criteria:

* Any individual present during the community events at the "five points" (barbershop, hair/beauty salon store or salon, corner store/grocery/neighborhood restaurant, laundromats, car service provider [e.g. gas station, mechanic, car wash]) in predominantly Black communities in Miami where HIV prevalence is high.
* Pre- and Post-assessment: Individuals are only eligible to complete the survey one time during the Pre-Intervention and during the Post-Intervention phases.
* Intervention: Individuals are only eligible to participate in the Intervention phase of this study once every 6 months.

Exclusion Criteria:

* Individuals who are unable to completely and fully understand the informed (verbal) consent process and the study procedures.
* Individuals who have previously completed the survey during the Pre-Intervention and Post-Intervention phases.
* Individuals who have participated in the Intervention phase of this study within less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20400 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in number of residents with recent HIV testing | Up to 23 months
  Will be reported as proportion of residents with recent (within 12 months) HIV testing as measured by Five Point Initiative - Community Survey
Change in number of residents with PrEP prescription | Up to 23 months
  Will be reported as proportion of residents with PrEP prescription as measured by Five Point Initiative - Community Survey
Change in PrEP knowledge as measured by Five Point Initiative - Community Survey | Baseline and up to 23 months
  Will be reported as the proportion of residents that indicated 'Yes' on the survey.

SECONDARY OUTCOMES:
Change in condom use as measured by Five Point Initiative - Community Survey | Baseline and up to 23 months
  Will be reported as the proportion of residents that indicated 'No' on the survey
Change in condom access as measured by Five Point Initiative - Community Survey | Baseline and up to 23 months
  Will be reported as the proportion of residents that indicated 'Yes' on the survey
Proportion of residents with recent HIV testing by health organizations | Up to 23 months
  Proportion of residents with recent (within 12 months) HIV testing by each of the participating health organizations.
Number of residents with PrEP prescription by health organizations | Up to 23 months
  Number of residents with PrEP prescription by each of the participating health organizations.

CONTACTS AND LOCATIONS:
Overall Officials: Sannisha Dale, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No